CLINICAL TRIAL: NCT04759209
Title: Development and Validation of a Machine Learning Based Virtual Biopsy System in Kidney Transplant Patients
Brief Title: Development and Validation of a Virtual Biopsy System in Kidney Transplant
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Collaborators: Mayo Clinic (Other); KU Leuven (Other); University of Liege (Other); University of British Columbia (Other); Hospital Clinic of Barcelona (Other); Assistance Publique - Hôpitaux de Paris (Other); Hospital Vall d'Hebron (Other); Hospital Universitari de Bellvitge (Other); Clinical Hospital Centre Zagreb (Other); University of Alberta (Other); University of Adelaide (Other)
Responsible Party: Sponsor
Other Study IDs: VirtualBx/KT
Record Dates: First submitted 2021-02-11; First posted 2021-02-18 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Day-zero biopsy; Machine learning; Non-invasive biopsy; Common parameters
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biopsies

SUMMARY:
Currently, kidney allograft biopsies are routinely performed to determine diagnosis and prognosis of kidney allografts. The histological interpretation of these biopsies is based on the Banff consensus for renal allograft pathology. The purpose of this study is to provide to the physicians a reliable estimation of renal allograft lesions of the day zero biopsy (kidney donor biopsy performed before transplantation).

DETAILED DESCRIPTION:
In kidney transplantation, day-zero biopsies are essential to assess organ quality and discriminate the donor transmitted or acquired lesions and disease progression post-transplant. However, many centers worldwide do not perform those biopsies because they are invasive and costly. We aimed to develop and validate a non-invasive virtual biopsy system. Our goal was to provide clinicians with a virtual biopsy system to guide diagnostics, therapeutics and immediate patient management post-transplant and to minimize additional risks and costs to perform day-zero biopsies only using standard donor parameters. To circumvent these limitations, we sought to build and validate a virtual biopsy system that uses routinely collected donor parameters to predict kidney day-zero biopsy results. Since machine learning has demonstrated its clinical relevance in many medical specialties and superior performance to logistic regression, we based our analyses on machine learning methods as well as traditional statistical approaches using large and qualified international cohort donors who underwent routine and protocolized collection of donor parameters together with day-zero biopsy assessment using the standards of the international Banff allograft histopathology classification.

ELIGIBILITY:
Inclusion Criteria:

- Kidney donors who underwent kidney biopsies performed prior to kidney transplantation, aged at least 18 years old.

Exclusion Criteria:

* inadequate biopsies according to Banff international classification (number of glomeruli less than 10),
* biopsies with two or more Banff scores of interest missing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living or deceased kidney donors who underwent a kidney biopsy performed prior to kidney transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 12992 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Arteriosclerosis score according to Banff International Classification | up to 1 day post-transplant
  Arteriosclerosis defined by arterial intimal thickening in the most severely affected artery (Banff "cv" score)
Arteriolar Hyalinosis score according to Banff International Classification | up to 1 day post-transplant
  arteriolar hyalinosis defined by periodic acid-Schiff (PAS)-positive arteriolar hyaline thickening (Banff "ah" score),
Interstitial fibrosis and tubular atrophy score according to Banff International Classification | up to 1 day post-transplant
  interstitial fibrosis and tubular atrophy computed with the extent of cortical fibrosis (Banff "ci" score) and cortical tubular atrophy (Banff "ct" score).
Continuous percentage of sclerotic glomeruli | up to 1 day post-transplant
  continuous percentage of sclerotic glomeruli is defined by the percentage of the total number of glomeruli affected by global sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, Principal Investigator — Paris Translational Research Center for Organ Transplantation
Locations (1):
- Paris Transplant Group, Paris, France

IPD SHARING:
Plan to Share IPD: No